CLINICAL TRIAL: NCT05245669
Title: A Randomized, Double-blind, Three-arm, Parallel-group, Single-dose Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety, Tolerability, and Immunogenicity of Denosumab (ENZ215, EU-sourced Prolia®, and US-sourced Prolia®) in Healthy Adult Male Volunteers
Brief Title: Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety, Tolerability, and Immunogenicity of Biosimilar Denosumab With Prolia® in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enzene Biosciences Ltd. (Industry)
Collaborators: Alkem Laboratories Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALK22/ENZ215-DEN1; 2021-004177-32 (EudraCT Number)
Record Dates: First submitted 2022-01-11; First posted 2022-02-18 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Intervention Model Description: Arm 1: ENZ215 Arm 2 : EU Sourced Prolia Arm 3: US Sourced Prolia
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ENZ215 (Experimental): ENZ215 Injection:- 60 mg Denosumab (ENZ215) will be administered subcutaneously on day 1.
  Interventions: Biological: ENZ215
- EU Sourced Prolia (Active Comparator): EU sourced Prolia Injection:- 60 mg Denosumab (EU sourced Prolia) will be administered subcutaneously on day 1.
  Interventions: Biological: EU Sourced Prolia
- US Sourced Prolia (Active Comparator): US sourced Prolia Injection:- 60 mg Denosumab (US sourced Prolia) will be administered subcutaneously on day 1.
  Interventions: Biological: US Sourced Prolia

INTERVENTIONS:
Biological: ENZ215 — healthy volunteers receive ENZ215 (60mg) once
  Arms: ENZ215
Biological: EU Sourced Prolia — healthy volunteers receive Denosumab (60mg) once
  Arms: EU Sourced Prolia
Biological: US Sourced Prolia — healthy volunteers receive Denosumab (60mg) once
  Arms: US Sourced Prolia

SUMMARY:
This is a randomized, double-blind, three-arm, parallel-group, single-dose study to demonstrate bioequivalence of ENZ215 and EU- and US-sourced Prolia after a single 60-mg dose administered subcutaneously in healthy adult male volunteers.

DETAILED DESCRIPTION:
Approximately 207 subjects will be enrolled into 3 groups (69 in each group) in parallel. The subjects may be enrolled in multiple groups at the site. All eligible subjects will be assigned to one of the three treatment groups in 1:1:1 ratio i.e. ENZ215 or US-sourced Prolia® or EU-sourced Prolia® to enter into the study period of 39 weeks. The study duration will be approximately 16 months (i.e. 6 months of recruitment period, 4 weeks of screening period and approximately 39 weeks (270 days) of study period).

Each subject will be required to visit the site for a total of 20 visits: visit 1 - screening visit, visit 2 - day 0 to day 2, visit 3 - day 3, visit 4 - day 4, visit 5 - day 5, visit 6 - day 6, visit 7 - day 8, visit 8 - day 10, visit 9 - day 12, visit 10 - day 16, visit 11 - day 21, visit 12 - day 28 (week 4), visit 13 - day 42 (week 6), visit 14 - day 63 (week 9), visit 15 - day 90 (week 13), visit 16 - day 119 (week 17), visit 17 - day 147 (week 21), visit 18 - day 180 (week 26), visit 19 day - 224 (week 32), and visit 20 - day 270 (week 39). A window period of ±1 day is allowed for visit 12 (day 28), window period of ±3 days are allowed from day 42 (week 6) to day 180 (week 26), A window period of ±5 days are allowed from day 224 (week 32) to day 270 (week 39).

End of Study Assessment will be performed on day 270 (week 39) or at the time of early discontinuation of the subject.

ELIGIBILITY:
INCLUSION CRITERIA

The subjects will be included in the study based on the following criteria:

1. Able to understand and give written, voluntary informed consent for the study
2. Healthy adult male volunteers between 28 to 55 years of age (both inclusive)
3. Body Mass Index (BMI) ≥ 18.50 and ≤ 30.00 kg/m2 at the time of screening
4. Medically healthy with no clinically significant medical history, vital signs, physical examination, and laboratory profiles
5. Normal or clinically acceptable 12-lead electrocardiogram, QT interval corrected for heart rate (QTc interval)* ≤ 450 msec at the time of screening
6. Subjects with negative alcohol test (breath analyzer or any suitable test) at the time of screening and admission (pre-dose)
7. Male subjects with female partners who agree to use effective contraception during study#
8. Male subjects who agree not to donate sperm during study
9. Willing and able to comply with the protocol requirements
10. Willing for multiple sampling and admission at the phase 1 study site day before dosing.

    * Note: QTc interval will be calculated using the Bazette and Fridericia formula.

      * Effective contraception: A non-vasectomised Male volunteers with female partners of child bearing potential should use dual method of contraception i.e. condom with spermicide method of contraception.

Female partners should use hormonal or non-hormonal method of contraception. (No restrictions are required for a vasectomised male provided his vasectomy has been performed 4 months or more prior to the first dosing. A male who has been vasectomised less than 4 months prior to the first dosing must follow the same restrictions as a non-vasectomised male).

EXCLUSION CRITERIA

The subjects will be excluded from the study based on the following criteria:

1. Known hypersensitivity to Denosumab or to any of the components of the study drug
2. Participating or has received any investigational drug (or is currently using an investigational device) within 30 days before receiving the study drug, or at least 10 times the respective elimination halflife (whichever period is longer) *

   * For monoclonal antibody refer exclusion criteria number 18 and 19
3. A serious infection (associated with housing and/or required intravenous anti-infectives) within 6 months before study drug administration and/or any active infection within 4 weeks of screening requiring oral or systemic antibiotics
4. History of significant drug abuse within 12 months before screening or a use of soft drugs (such as marijuana) within 3 months before the screening visit or hard drugs (such as cocaine, phencyclidine, and crack etc.) within 12 months before screening
5. Smokers who smoke ≥ 10 cigarettes or equivalent per day within 90 days prior to screening
6. Subjects with positive urine screen for drugs of abuse at the time of screening or check-in
7. Subjects with Urine Cotinine > 500ng/ml at the time of screening or check-in
8. Subjects with risk of osteonecrosis of the jaw i.e. poor oral hygiene, periodontal disease, poorly fitting dentures, history of dental disease or have undergone invasive dental procedures e.g. tooth extractions within last 6 months prior to screening.
9. Subjects with a predictable risk of invasive dental surgery during the 9 months after dosing or with planned invasive dental procedure
10. Subjects with known bone disease or recent fracture or abnormalities of calcium metabolism
11. Loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL within 30 days, or more than 499 mL within 56 days before dosing
12. History of immunodeficiency (including those subjects with a positive test for human immunodeficiency virus [HIV] at screening)
13. Have a positive result for hepatitis B antigen test (HBsAg) or hepatitis C antibody test (HCAb), or show evidence of possible infection
14. Major surgical procedure within 28 days of dose of investigational product.
15. Male subjects having pregnant female partner at the time of screening.
16. Subject with a history of recurrent or chronic infections
17. Received live vaccines within 4 weeks or who may require live vaccine(s) during the study duration
18. Prior use of denosumab
19. Have previously been exposed to a monoclonal antibody or fusion protein within 270 days (other than denosumab) prior to randomisation and/or there is confirmed evidence or clinical suspicion of immunogenicity from previous exposure to a monoclonal antibody or fusion protein.
20. Any reason/condition which would preclude subject's participation in the study as per the Investigator's opinion or warnings and contraindications in the prescribing information of Prolia
21. Subjects with suspected signs and symptoms of COVID-19/confirmed novel coronavirus infection (COVID-19).

Ages: 28 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy adult male of age 28-55 years
Enrollment: 207 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nadine Abdullah, Principal Investigator — Celerion GB Ltd.
Locations (2):
- MC Comac Medical, Sofia, Sofia City Province, Bulgaria
- MTZ Clinical Research powered by Pratia, Pratia S.A, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ENZ215 | EU Sourced Prolia | US Sourced Prolia
Started | 68 | 69 | 70
Completed | 66 | 67 | 67
Not Completed | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Participants were healthy adult male volunteers between 28 to 55 years of age.
Groups:
- ENZ215: ENZ215 is the proposed biosimilar for Prolia® (denosumab). Subjects in this arm received a single 60 mg dose of ENZ215 as a subcutaneous injection.
  ENZ215 (denosumab biosimilar) : Single dose of 60mg SC administered
- EU Sourced Prolia: EU-Prolia® (denosumab) is the proposed active comparator for ENZ215. Subjects in this arm received a single 60 mg dose of EU-Prolia® as a subcutaneous injection.
  EU-Prolia® : Single dose of 60mg SC administered
- US Licensed Prolia: US-Prolia® (denosumab) is the proposed active comparator for ENZ215. Subjects in this arm received a single 60 mg dose of US-Prolia® as a subcutaneous injection.
  US-Prolia® : Single dose of 60mg SC administered
- Total: Total of all reporting groups
Arm/Group | ENZ215 | EU Sourced Prolia | US Licensed Prolia | Total
Number analyzed (Participants) | 68 | 69 | 70 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (8.1) | 38.9 (7.7) | 40.1 (7.8) | 39.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 68 | 69 | 70 | 207
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 0 | 1
  White | 67 | 69 | 70 | 206
Height [Mean (Standard Deviation); unit: cm] | 178.39 (6.22) | 178.96 (6.44) | 178.41 (7.69) | 178.59 (6.79)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.219 (2.601) | 26.260 (2.760) | 25.562 (2.835) | 26.010 (2.740)
Weight [Mean (Standard Deviation); unit: kg] | 83.62 (10.75) | 84.16 (10.34) | 81.56 (11.67) | 83.10 (10.94)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Drug Concentration (Cmax) of ENZ215 and EU- and US-sourced Prolia®
Description: A total of twenty four blood PK samples of 2.5 mL each were collected from each subject in the study. Pre-dose sample were collected within 30 minutes prior to IP administration. Post-dose samples up to Day 2 were collected within ± 10 minutes, within ± 2 hours from Day 3 to Day 21, within ± 1 day on Day 28, within ± 3 days from Day 42 to Day 180 and within ±5 days from Day 224 to Day 270.
  Serum concentrations of denosumab were measured at central laboratory by a validated analytical method.
Time Frame: 270 days
Population: Pharmacokinetic population includes subjects who complied sufficiently with the protocol, who received a single-dose of the study drug and had 1 pre-dose and at least 1 post-dose measurement of any of the PK assessment not impacted by any protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | ENZ215 | EU Sourced Prolia | US Licensed Prolia
Number analyzed (Participants) | 68 | 69 | 69
ng/ml | 7662.99 (32.6) | 7742.64 (23.2) | 8033.14 (24.9)

2. Primary Outcome: Area Under the Drug Concentration-time Curve From Day 0 to Day 270 (AUC0-t) of ENZ215, EU- and US-sourced Prolia®. and EU- and US-sourced Prolia®
Description: as for outcome 1
Time Frame: 270 days
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | ENZ215 | EU Sourced Prolia | US Licensed Prolia
Number analyzed (Participants) | 68 | 69 | 69
h*ng/mL | 7508134.18 (36.8) | 7674912.81 (24.9) | 7842297.13 (28.8)

3. Primary Outcome: Area Under the Drug Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of ENZ215, EU- and US-sourced Prolia®. and EU- and US-sourced Prolia®
Description: as for outcome 1
Time Frame: 270 days
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | ENZ215 | EU Sourced Prolia | US Sourced Prolia
Number analyzed (Participants) | 68 | 69 | 69
h*ng/mL | 7622698.42 (36.4) | 7779487.60 (24.7) | 7934699.65 (28.9)

4. Secondary Outcome: Partial Area Under the Drug Concentration-time Curve From Time 0 (Pre-dose) to Day 28
Description: AUC0-28 days were compared between ENZ215 and Prolia® using tests after log-transformation wherever appropriate.
Time Frame: 28 days
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | ENZ215 | EU Sourced Prolia | US Sourced Prolia
Number analyzed (Participants) | 66 | 67 | 67
h*ng/mL | 3608894.44 (28.9) | 3721138.61 (20.6) | 3796048.41 (22.5)

5. Secondary Outcome: Time to Reach Cmax (Tmax)
Description: The non-parametric analysis was used for the comparison of tmax between ENZ215 and Prolia®.
Time Frame: 270 days
Measure: Median (Full Range); unit: hours
Arm/Group | ENZ215 | EU Sourced Prolia | US Sourced Prolia
Number analyzed (Participants) | 68 | 69 | 69
hours | 120.62 [47.22 to 360.63] | 120.08 [46.93 to 359.75] | 120.28 [46.98 to 479.92]

6. Secondary Outcome: Terminal Elimination Half-life (t1/2)
Description: t1/2 was compared between ENZ215 and Prolia® using tests after log-transformation wherever appropriate.
Time Frame: 270 days
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ENZ215 | EU Sourced Prolia | US Sourced Prolia
Number analyzed (Participants) | 66 | 67 | 67
hours | 450.745 (28.3) | 450.207 (23.2) | 441.262 (27.1)

7. Secondary Outcome: Apparent Systemic Clearance (CL/F)
Description: CL/F was compared between ENZ215 and Prolia® using tests after log-transformation wherever appropriate.
Time Frame: 270 days
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | ENZ215 | EU Sourced Prolia | US Sourced Prolia
Number analyzed (Participants) | 66 | 67 | 67
mL/h | 0.008 (36.4) | 0.008 (24.7) | 0.008 (28.9)

8. Secondary Outcome: Area Under the Effect Curve (AUEC) From Time 0 to Day 270 for Serum CTX-1 Percent Inhibition Percent Inhibition
Description: The AUEC was calculated as the area under the effect curve from baseline until CTX-1 values return to baseline for the first time.
  A total of sixteen (16) blood samples for serum CTX-1 estimation of 3.5 mL each was collected from each subject in the study. For CTX-1, blood samples were collected at the same time and after a minimum of 10 hours of fasting.
Time Frame: 270 days
Population: Pharmacodynamic population includes subjects who complied sufficiently with the protocol, who received a single-dose of the study drug and had 1 pre-dose and at least 1 post-dose measurement of any of the PD assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*%
Arm/Group | ENZ215 | EU Sourced Prolia | US Sourced Prolia
Number analyzed (Participants) | 68 | 69 | 69
h*% | 432174.780 (20.1) | 442806.204 (13.6) | 436622.000 (18.6)

9. Other Pre Specified Outcome: Number of Subjects Who Developed Denosumab Neutralizing Antibodies and Antidrug Antibodies. Antibodies
Description: A total of 10 blood Immunogenicity assessment samples of 5.0 mL for NAb and ADA were collected from each subject in the study.
  The frequency and percentage of positive ADA or NAb result was provided. The proportion of positive ADA or NAb in each treatment group was compared using chi-square or Fisher's exact tests. The p-value, relative risk, and corresponding 95% CI was presented.
Time Frame: 270 days
Population: Total 207 subjects randomized i.e. in 68 subjects in ENZ215, 70 subjects in US-Prolia® & 69 subjects in EU-Prolia® randomized. However, in US-Prolia® 69 subjects dosed as 1 subject withdrawn his consent before dosing, in ENZ215 & EU-Prolia® all randomized subjects dosed. Hence in US-Prolia® 69 subjects, EU-Prolia® 69 subjects & ENZ215 68 subjects evaluated in the study.
  Number subjects showed nAb.
Measure: Number; unit: participants
Arm/Group | ENZ215 | EU Sourced Prolia | US Sourced Prolia
Number analyzed (Participants) | 68 | 69 | 69
participants
  ADA positive subjects | 68 | 69 | 69
  nAb positive subjects | 3 | 3 | 2

10. Other Pre Specified Outcome: Incidence of Adverse Events
Description: Adverse events and SAEs as and when occurred, were properly recorded, evaluated, managed, and reported from signing informed consent till end of Study Assessment visit. All AEs were summarized using appropriate medical coding dictionary.
Time Frame: 270 days
Population: Total 207 subjects randomized i.e. in 68 subjects in ENZ215, 70 subjects in US-Prolia® & 69 subjects in EU-Prolia® randomized. However, in US-Prolia® 69 subjects dosed as 1 subject withdrawn his consent before dosing, in ENZ215 & EU-Prolia® all randomized subjects dosed. Hence in US-Prolia® 69 subjects, EU-Prolia® 69 subjects & ENZ215 68 subjects evaluated in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | ENZ215 | EU Sourced Prolia | US Sourced Prolia
Number analyzed (Participants) | 68 | 69 | 69
Participants | 28 | 39 | 32

ADVERSE EVENTS:
Time Frame: from signing of informed consent to 270 days that is end of study
Description: All AEs were classified according to the Medical Dictionary for Regulatory Activities (MedDRA), Version 25.0 for subjects of site 01 and from MedDRA dictionary, Version 26.1 for subjects of site 02 and 03.
Groups:
- EU Sourced Prolia®: EU-Prolia® (denosumab) is the proposed active comparator for ENZ215. Subjects in this arm received a single 60 mg dose of EU-Prolia® as a subcutaneous injection.
  EU-Prolia® : Single dose of 60mg SC administered
- US Licensed Prolia®: US-Prolia® (denosumab) is the proposed active comparator for ENZ215. Subjects in this arm received a single 60 mg dose of US-Prolia® as a subcutaneous injection.
  US-Prolia® : Single dose of 60mg SC administered.
Arm/Group | ENZ215 | EU Sourced Prolia® | US Licensed Prolia®
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/68 | 1/69 | 0/69
Other Adverse Events (participants affected / at risk) | 28/68 | 39/69 | 32/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENZ215 (N=68) | EU Sourced Prolia® (N=69) | US Licensed Prolia® (N=69)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENZ215 (N=68) | EU Sourced Prolia® (N=69) | US Licensed Prolia® (N=69)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 7 (7) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 6 (6) | 1 (1)
Headache (Nervous system disorders) | 9 (18) | 9 (11) | 14 (20)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 11 (13) | 13 (14)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Migraine (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT05245669/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT05245669/SAP_001.pdf